CLINICAL TRIAL: NCT04503694
Title: A Phase II Trial of Neoadjuvant Regorafenib in Combination with Nivolumab and Short-course Radiotherapy in Stage II-III Rectal Cancer
Brief Title: Neoadjuvant Regorafenib in Combination with Nivolumab and Short-course Radiotherapy in Stage II-III Rectal Cancer
Acronym: REGINA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-REGINA-2020; 2024-516554-22-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-28; First posted 2020-08-07 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer Stage II; Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms | interventions — Nivolumab; regorafenib; Tablets; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): * Induction treatment: treatment with nivolumab (240 mg intravenously on day 1 and 14) and regorafenib (60 mg/day orally from day 1 to 14)
  * Standard SCRT: consists of 25 Gy delivered in 5 fractions (from day 22 to 26)
  * Consolidation treatment: treatment with nivolumab (240 mg intravenously on day 29, 43 and 57) and regorafenib (60 mg/day orally from day 29 to 49)
  * Surgery: Surgical resection will be performed according to the principles of TME (between day 74 and 87, i.e., between 7 to 8 weeks after completion of SCRT). As an alternative to surgery, subjects who achieve cCR can be offered a watch & wait approach.
  * Adjuvant chemotherapy: Administration of adjuvant chemotherapy will be left to the discretion of the treating physician The study also includes translational procedures (collection of tumour biopsies, blood and stool samples at pre-specified time points) for exploratory molecular and immune contexture analyses. These are mandatory for all study subjects.
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution; Drug: Regorafenib 30 MG Oral Tablet; Radiation: Radiotherapy; Procedure: Surgery; Procedure: Non-operative Management

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML Intravenous Solution — Nivolumab will be given at a dose of 240 mg during the pre-operative phase only as indicated below:
  * On day 1 and 15, during the "Induction treatment"
  * On day 29, 43 and 57, during the "Consolidation treatment"
Drug: Regorafenib 30 MG Oral Tablet — Regorafenib will be administered orally once a day at a dose of 60 mg/day (2 tablets of 40 mg), during the pre-operative phase only as indicated below:
  * From day 1 to 14, during the "Induction treatment"
  * From day 29 to 49, during the "Consolidation treatment"
Radiation: Radiotherapy — All study subjects will receive 5 daily fractions of radiotherapy. Each fraction will consist of 5 Gy for a total dose of 25 Gy. Radiotherapy is to start on day 22 and to finish on day 26.
Procedure: Surgery — Subject will undergo surgical resection of the primary tumour in the rectum between day 74 and 87. Surgery must be performed according to the principles of total mesorectal excision as described by Heald et al. The type of surgical approach (low anterior resection or abdominoperineal resection, etc.) will be left to the discretion of the treating surgeon.
Procedure: Non-operative Management — Subjects who achieve cCR after pre-operative treatment can, after discussion with the local investigator, decline surgery and opt for a non-operative management. cCR will need to be confirmed between day 67 and 74 by the following procedures per local practise:
  * Digital rectal examination
  * Rectal endoscopy
  * Rectal MRI Subjects who achieve near cCR at the first assessment time point after pre-operative treatment, can be re-assessed 6 to 8 weeks later with the same procedures. If cCR is diagnosed, they can opt for watch & wait, otherwise they would need to undergo surgical resection.
  Subjects who opt for a non-operative management will be followed for tumour recurrence and survival for 5 years after end of treatment visit. Follow-up for these subjects will be more intensive than that for subjects undergoing surgery

SUMMARY:
This is a multicenter, single-arm, phase II study of nivolumab in combination with regorafenib in subjects with locally-advanced rectal cancer who are eligible for a curative treatment including pre-operative SCRT and TME(or watch & wait approach). The study is based on the Simon's two-stage design and a maximum of 60 subjects will be enrolled. In addition to the standard efficacy interim analysis according to the statistical design, a safety interim analysis will be performed on the first 6 subjects who have completed the study treatment to ensure safe continuation of the study investigation.

Eligible subjects will be treated according to the following sequential treatment plan:

* Induction treatment: This consists of treatment with nivolumab (240 mg intravenously, on day 1 and 15) and regorafenib (60 mg/day orally, from day 1 to 14)
* Standard SCRT: This consists of 25 Gy delivered in 5 fractions (from day 22 to 26)
* Consolidation treatment: This consists of treatment with nivolumab (240 mg intravenously, on day 29, 43 and 57) and regorafenib (60 mg/day orally, from day 29 to 49)
* Surgery: Surgical resection will be performed according to the principles of TME (between day 74 and 87, i.e., between 7 to 8 weeks after completion of SCRT). As an alternative to surgery, subjects who achieve cCR can be offered a watch & wait approach.
* Adjuvant chemotherapy: Administration of adjuvant chemotherapy will be left to the discretion of the treating physician

The study also includes translational procedures (i.e. collection of tumour biopsies, blood samples and stool samples at pre-specified time points) for exploratory molecular and immune contexture analyses. These are mandatory for all study subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male
2. Age ≥ 18 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. Histologically or cytologically verified adenocarcinoma of the rectum
5. Tumour with distal border below the peritoneal reflection and within 15 cm from the anal verge
6. Stage cT3/T4a and Nany or cT1-2 and N+ as documented by baseline pelvic MRI
7. Absence of distant metastases as shown by baseline computed tomography (CT) of the thorax-abdomen or CT scan of the thorax and MRI of the abdomen
8. Adequate haematological function as defined by absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count ≥100 × 109/L, and haemoglobin ≥9 g/dL
9. Adequate hepatic function as defined by a total bilirubin level ≤1.5 × the upper limit of normal (ULN) range (excluding subjects with known Gilbert's syndrome) and alanine aminotransferase (ALT) levels ≤2.5 × ULN
10. Adequate renal function as defined by an estimated creatinine clearance ≥30 mL/min according to the Cockcroft-Gault or Wright formula
11. Negative serum pregnancy test at screening (up to 7 days before treatment start) for women of childbearing potential
12. Women of childbearing potential must agree to use of one highly effective method of contraception prior study entry, during the course of the study and at least 5 months after the last administration of study treatment.
13. Men with childbearing potential partner must agree to use condom during the course of this study and for at least 5 months after the last administration of the study treatment.
14. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
15. Absence of clinical conditions that, in the opinion of the investigator, would contraindicate neoadjuvant therapy and/or surgery
16. Life expectancy of at least 3 months
17. Completion of all necessary screening procedures within 28 days prior to enrolment.
18. Signed Informed Consent form (ICF) obtained prior to any study related procedure.

Exclusion Criteria:

1. Any prior or concurrent surgery, chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for rectal cancer. Concurrent use of hormones for noncancer-related conditions (i.e., insulin for diabetes and hormone replacement therapy) is acceptable.
2. Any contraindication to pelvic irradiation as evaluated by the investigator
3. Prior organ transplantation, including allogeneic stem cell transplantation
4. Clinically significant acute or chronic infections including, among others:

   * known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
   * known history of testing positive for hepatitis B virus (HBV) surface antigen or anti-hepatitis C virus (HCV) antibody and confirmatory HCV ribonucleic acid (RNA) test
5. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent (subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible)
6. Systemic corticosteroids administered as hormone replacement or as immunosuppressants at doses exceeding 10 mg/day of prednisone or equivalent. Other immunosuppressive medications including, but not limited to methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of treatment-related AEs or in subjects with contrast allergies is acceptable. A temporary period of steroids is allowed for different indications, at the discretion of the investigator (i.e., chronic obstructive pulmonary disease, radiation, nausea, etc.). Administration of steroids through a route known to result in a minimal systemic exposure [topical, intranasal, intro-ocular, or inhalation] is acceptable.
7. Known severe hypersensitivity reactions to the investigational treatments, or any excipients or non-investigational medicinal products or concomitant medications
8. Pregnant and/or lactating women
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure, uncontrolled arterial hypertension, or serious cardiac arrhythmia requiring medication
10. Prior myocarditis
11. Known history of immune colitis, immune pneumonitis, pulmonary fibrosis or other medical conditions (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment
12. Vaccination within 28 days of the first dose of study treatment and while on trial (except for administration of inactivated vaccines)
13. Other invasive malignancy within 2 years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured. Anti-neoplastic treatment received in the past for malignancies cured 2 or more years before enrolment are permitted.
14. Any investigational anti-cancer therapy other than the protocol specified therapies.
15. Strong inhibitors of CYP3A4 activity (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin and voriconazole), strong UGT1A9 inhibitors (e.g. mefenamic acid, diflunisal, and niflumic acid), and strong inducers of CYP3A4 (e.g. rifampicin, phenytoin, carbamazepine, phenobarbital and St. John's wort) from 28 days before study enrolment up to the end of study treatment.
16. Major surgery within 28 days of the first dose of study treatment
17. Presence of gastrointenstinal perforation of fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of the combination of nivolumab and regorafenib when administered before and after standard, pre-operative short-course radiation therapy. | immediately after the surgery
  Measurement of the clinical (cCR) and pathological complete response (pCR) rate in subjects with pMMR/MSS tumours This will be evaluated in the mITT population and defined as the absence of viable tumour cells in the surgical specimens.
  Rate of pCR will be presented as number of subjects and percentage, along with a 95% confidence interval.

SECONDARY OUTCOMES:
Assessment of the toxicity according to the NCI CTCAE version 5.0. | 5 months after the last administration of study treatment
  The type, frequency and severity of adverse events will be analysed in the mITT population.
Assessment of the proportion of subjects who complete systemic treatment, radiotherapy and surgery according (if perfomed) to the study protocol. | immediately after the surgery (if performed)
  This is will be evaluated in the Intention to Treat (ITT) population to assess the feasibility of combining regorafenib with nivolumab in the setting of locally-advanced rectal cancer as demonstrated by subject compliance with the investigational strategy, SCRT and surgery (if performed)
Evaluation of the efficacy of the combination of nivolumab and regorafenib when administered before and after standard, pre-operative short-course radiation therapy. | immediately after the surgery (if performed)
  RO resection rate will be analysed in the mITT population and defined as the proportion of subjects who undergo surgical resection of the tumour with clear margins (i.e., >1 mm).
Evaluation of the immune activation induced by the investigational treatment regorafenib with nivolumab | Before (biopsy at week 3) and immediately after surgery (surgical specimen) (if performed)
  CD3 and CD8 T-cells infiltrate increase in post-treatment tumour tissue samples
Evaluation of the efficacy of the combination of nivolumab and regorafenib when administered before and after standard, pre-operative short-course radiation therapy. | immediately after the surgery (if performed)
  The rate of complete/near complete pathological tumour regression will be evaluated in the mITT population and defined as the proportion of subjects who achieve pathological tumour regression grade (pTRG) 3 or 4 according to the Dworak pTRG score.
Evaluation of the efficacy of the combination of nivolumab and regorafenib when administered before and after standard, pre-operative short-course radiation therapy. | 5 years after end of treatment
  The Event-free survival (EFS) will be evaluated in the mITT population and calculated from the date of registration to the date of occurrence of any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause. Kaplan Meier methods will be used to calculate EFS rates along with 95% confidence intervals.
Evaluation of the efficacy of the combination of nivolumab and regorafenib when administered before and after standard, pre-operative short-course radiation therapy. | 5 years after end of treatment
  The Overall survival (OS) will be evaluated in the mITT population and calculated from the date of registration to the date of death from any cause. Kaplan Meier methods will be used to calculate OS rates along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sclafani, MD, Study Chair — Jules Bordet Institute
Locations (10):
- Belgium (10):
  - Institut Jules Bordet, Anderlecht
  - Erasme, Brussels
  - Chirec Delta, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZAntwerpen, Edegem
  - UZ Gent, Ghent
  - Grand Hopital de Charleroi, Gilly
  - AZ Groeninge, Kortrijk
  - CHU Ambroise Paré, Mons
  - CHR Namur, Namur

IPD SHARING:
Plan to Share IPD: Undecided